CLINICAL TRIAL: NCT03179761
Title: High vs. Standard Dose Flu Vaccine in Adult Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Natasha Halasa, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VICC CTT 1733; NCI-2017-00466 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic Cell Transplantation
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (HD-TIV) (Experimental): Patients received HD-TIV intramuscularly once at baseline (day 0) and again between 28-42 days later.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Trivalent Influenza Vaccine
- Group 2(SD-QIV) (Active Comparator): Patients received SD-QIV intramuscularly once at baseline (day 0) and again between 28-42 days later.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Quadrivalent Inactivated Influenza Vaccine — Standard Dose Quadrivalent Influenza Vaccine given intramuscularly
  Arms: Group 2(SD-QIV)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Trivalent Influenza Vaccine — High Dose Trivalent Influenza Vaccine given intramuscularly
  Arms: Group I (HD-TIV)

SUMMARY:
This randomized phase II studies the side effects of high-dose trivalent influenza vaccine or standard-dose quadrivalent inactivated influenza and how well they work in treating adult patients undergoing stem cell transplant. Season influenza can cause more severe infections in patients who have had a stem cell transplant since their immune system doesn't work as well. Influenza vaccine may provide better protection against flu in adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether high dose (HD)-trivalent influenza vaccine (TIV) compared with standard dose (SD)-quadrivalent inactivated influenza vaccine (QIV) will increase the probability of achieving a >= 4-fold rise in hemagglutination inhibition assay (HAI) titer, >= 1:40 HAI titer, or a higher geometric mean titer (GMT) titer to influenza A antigens in adult hematopoietic cell transplantation (HSCT) recipients.

SECONDARY OBJECTIVES:

I. To determine whether HD-TIV compared with SD-QIV will increase the probability of achieving a >= 4-fold rise in HAI titers, >= 1:40 HAI titer, or higher GMT titers to influenza B antigens in adult HSCT recipients.

II. To determine the frequency and severity of solicited local injection site adverse events (e.g. pain/tenderness, redness, and swelling at injection site) with HD-TIV compared to SD-QIV in adult HSCT recipients.

III. To determine the frequency and severity of solicited systemic adverse events (e.g. fevers, headache, fatigue/malaise, nausea, body ache/myalgia, general activity level, and vomiting) with HD-TIV compared to SD-QIV in adult HSCT recipients.

IV. To define the relationship between HAI titers, in vivo T and B cell phenotype, and in vitro influenza-specific T and B cell response in adult HSCT recipients receiving either HD-TIV or SD-QIV.

V. To correlate HAI responses to microneutralization responses. VI. To compare the persistent HAI and microneutralization assay (MN) titers for all four antigen seven months after the last vaccine dose to assess for persistence of antibody titers.

VII. To compare influenza detection by polymerase chain reaction (PCR) during influenza season in adult HSCT recipients receiving either HD-TIV or standard dose QIV.

OUTLINE: Patients are randomized into 1 of 2 groups.

GROUP I: Patients receive HD-TIV intramuscularly once at baseline and once between 28-42 days.

GROUP II: Patients receive SD-QIV intramuscularly once at baseline and once between 28-42 days.

After completion of study treatment, patients are contacted at 1-3 and 8-10 days after each vaccination visit.

ELIGIBILITY:
Inclusion criteria

1. Allogeneic HSCT recipients who are 3-23 months post-transplant;
2. ≥ 18 years of age;
3. Available for duration of study;
4. Patients with stable GVHD for at least 4 weeks will be eligible (stable is defined as no major change in systemic immunosuppressive therapy for worsening GVHD; adjustment of actual dose to obtain a stable target level is acceptable).
5. Can be reached by telephone and/or electronic communication
6. Subjects must have a platelet count of ≥30,000 to receive the immunizations. Patients requiring platelet transfusions are eligible to enroll and must have a platelet count ≥30,000 within 72 hours prior to their immunization, or platelet count ≥75,000 without transfusion documented within 30 days for subjects <12 months post- transplant and within 90 days for subjects 12-23 months post-transplant.

Exclusion criteria

1. History of hypersensitivity to previous influenza vaccination or severe hypersensitivity to eggs/egg protein;
2. History of Guillain-Barre syndrome;
3. Evidence of hematologic malignancy or disease relapse post-transplant (stable mixed chimerism is permitted);
4. History of receiving current seasonal influenza vaccine post-transplant;
5. Pregnant female;
6. History of proven influenza disease after September 1, 2018 prior to enrollment;
7. Non-allogeneic (e.g. autologous) or syngeneic hematopoietic SCT recipients;
8. History of known active infection with HIV
9. History of cirrhosis
10. History of known latex hypersensitivity;
11. Subjects who have received stem cell boost or delayed donor lymphocyte infusion within 90 days of enrollment, including day of enrollment
12. Receipt of. IVIG/SCIG <28 days prior to vaccination

Criteria for temporarily delaying vaccine administration: The following conditions are temporary or self-limiting, and a subject may be included in the study once the condition has resolved, provided that the subject is otherwise eligible:

1. Fever ≥100.4ºF/38.0ºC (oral measurement), or an acute illness within 48 hours of enrollment
2. Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks prior to potential study vaccination.

Note: if patients were eligible for vaccine 1, they will be eligible to receive vaccine 2 regardless of any changes on their GVHD status, unless it is deemed not medically safe to receive influenza vaccine.

For subjects who were enrolled and vaccinated in 2017-18, and 2018-19, the goal is to enroll these same subjects who participated the previous influenza season year and then administer the same vaccination as the previous year. These subjects are referred to as repeaters. For example, subjects enrolled in 2017-18 year were eligible to enroll again in 2018-19 as repeaters. For subjects enrolled in 2018-19 year and received at least one vaccine, will be eligible to be enrolled as repeaters for 2019-2020 season.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 138 adults were targeted with the expectation of a 20% drop out rate, as described in Section C17 in the protocol. We were able to enroll 124 subjects with a 15% dropout rate between Visit 1 and Visit 4.
Groups:
- Group 2 (SD-QIV): Patients received SD-QIV intramuscularly once at baseline (day 0) and again between 28-42 days later.
  Quadrivalent Inactivated Influenza Vaccine: Standard Dose Quadrivalent Influenza Vaccine given intramuscularly
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Started | 60 | 64
Visit 1 (Study vaccine was administered.) | 60 | 64
Visit 2 (Study vaccine was administered.) | 59 | 59
Visit 3 | 59 | 59
Visit 4 | 54 | 51
Visit 1 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment, and the study vaccine was administered. See protocol for criteria.) | 23 | 20
Visit 2 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment, and the study vaccine was administered. See protocol for criteria.) | 21 | 20
Visit 3 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment. See protocol for criteria.) | 19 | 20
Visit 4 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment. See protocol for criteria.) | 12 | 12
Completed (This includes subjects who completed all four visits for their first year of enrollment. This does not account for those who participated in a "repeater" year.) | 54 | 51
Not Completed | 6 | 13
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Investigator Request | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of their assigned vaccine
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV) | Total
Number analyzed (Participants) | 60 | 64 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 43 | 96
  >=65 years | 7 | 21 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.657 [34.448 to 61.643] | 59.986 [51.397 to 66.943] | 57.815 [42.358 to 64.101]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 34 | 42 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 58 | 62 | 120
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 3 | 8
  White | 51 | 60 | 111
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 64 | 124

OUTCOME MEASURES:

1. Primary Outcome: HD-TIV Compared With SD-QIV (Influenza A) - Immunogenicity
Description: Point estimates and 95% confidence intervals for proportion of subjects achieving seroprotection (≥1:40 HAI titer) and seroconversion (4-fold or greater rise in HAI titers from visit 1) for Influenza A antigens.
Time Frame: Visit 1 titers (baseline) were measured on day 0; visit 2 titers were measured 28-42 days after visit 1; visit 3 titers were measured 28-42 days after visit 2; and visit 4 titers were measured 138-222 days after visit 2.
Population: The number analyzed for each row represents the number of participants that completed the indicated visit and had a recorded HAI titer for the indicated antigen and visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Number analyzed (Participants) | 60 | 64
proportion of participants
  A/H1N1 Visit 2 GMT ≥1:40 | 0.62 [0.49 to 0.73] | 0.59 [0.46 to 0.70]
  A/H1N1 Visit 2 GMFR ≥ 4-Fold Rise | 0.23 [0.14 to 0.35] | 0.25 [0.16 to 0.37]
  A/H1N1 Visit 3 GMT ≥1:40: number analyzed (Participants) | 59 | 60
  A/H1N1 Visit 3 GMT ≥1:40 | 0.75 [0.63 to 0.84] | 0.73 [0.61 to 0.84]
  A/H1N1 Visit 3 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 59 | 60
  A/H1N1 Visit 3 GMFR ≥ 4-Fold Rise | 0.41 [0.29 to 0.53] | 0.39 [0.27 to 0.52]
  A/H1N1 Visit 4 GMT ≥1:40: number analyzed (Participants) | 57 | 56
  A/H1N1 Visit 4 GMT ≥1:40 | 0.66 [0.53 to 0.78] | 0.65 [0.51 to 0.78]
  A/H1N1 Visit 4 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 57 | 56
  A/H1N1 Visit 4 GMFR ≥ 4-Fold Rise | 0.34 [0.22 to 0.47] | 0.35 [0.22 to 0.49]
  A/H3N2 Visit 2 GMT ≥1:40 | 0.65 [0.52 to 0.76] | 0.60 [0.48 to 0.72]
  A/H3N2 Visit 2 GMFR ≥ 4-Fold Rise | 0.32 [0.21 to 0.44] | 0.19 [0.11 to 0.30]
  A/H3N2 Visit 3 GMT ≥1:40: number analyzed (Participants) | 59 | 60
  A/H3N2 Visit 3 GMT ≥1:40 | 0.78 [0.66 to 0.87] | 0.73 [0.61 to 0.84]
  A/H3N2 Visit 3 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 59 | 60
  A/H3N2 Visit 3 GMFR ≥ 4-Fold Rise | 0.49 [0.37 to 0.62] | 0.38 [0.26 to 0.51]
  A/H3N2 Visit 4 GMT ≥1:40: number analyzed (Participants) | 57 | 56
  A/H3N2 Visit 4 GMT ≥1:40 | 0.66 [0.53 to 0.78] | 0.49 [0.35 to 0.63]
  A/H3N2 Visit 4 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 57 | 56
  A/H3N2 Visit 4 GMFR ≥ 4-Fold Rise | 0.40 [0.27 to 0.53] | 0.27 [0.16 to 0.40]

2. Secondary Outcome: HD-TIV Compared With SD-QIV (Influenza B) - Immunogenicity
Description: Point estimates and 95% confidence intervals for proportion of subjects achieving seroprotection (≥1:40 HAI titer) and seroconversion (4-fold or greater rise in HAI titers from visit 1) for Influenza B antigens.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Number analyzed (Participants) | 60 | 64
proportion of participants
  B/Victoria Visit 2 GMT ≥1:40 | 0.73 [0.61 to 0.83] | 0.79 [0.68 to 0.88]
  B/Victoria Visit 2 GMFR ≥ 4-Fold Rise | 0.25 [0.15 to 0.37] | 0.17 [0.09 to 0.28]
  B/Victoria Visit 3 GMT ≥1:40: number analyzed (Participants) | 59 | 60
  B/Victoria Visit 3 GMT ≥1:40 | 0.92 [0.83 to 0.97] | 0.86 [0.75 to 0.93]
  B/Victoria Visit 3 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 59 | 60
  B/Victoria Visit 3 GMFR ≥ 4-Fold Rise | 0.44 [0.32 to 0.57] | 0.29 [0.18 to 0.41]
  B/Victoria Visit 4 GMT ≥1:40: number analyzed (Participants) | 57 | 56
  B/Victoria Visit 4 GMT ≥1:40 | 0.83 [0.71 to 0.91] | 0.73 [0.60 to 0.84]
  B/Victoria Visit 4 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 57 | 56
  B/Victoria Visit 4 GMFR ≥ 4-Fold Rise | 0.34 [0.22 to 0.47] | 0.18 [0.09 to 0.31]
  B/Yamagata Visit 2 GMT ≥1:40 | 0.72 [0.60 to 0.82] | 0.87 [0.78 to 0.94]
  B/Yamagata Visit 2 GMFR ≥ 4-Fold Rise | 0.07 [0.02 to 0.15] | 0.22 [0.13 to 0.33]
  B/Yamagata Visit 3 GMT ≥1:40: number analyzed (Participants) | 59 | 60
  B/Yamagata Visit 3 GMT ≥1:40 | 0.80 [0.68 to 0.89] | 0.88 [0.77 to 0.94]
  B/Yamagata Visit 3 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 59 | 60
  B/Yamagata Visit 3 GMFR ≥ 4-Fold Rise | 0.10 [0.04 to 0.20] | 0.27 [0.16 to 0.39]
  B/Yamagata Visit 4 GMT ≥1:40: number analyzed (Participants) | 57 | 56
  B/Yamagata Visit 4 GMT ≥1:40 | 0.64 [0.51 to 0.76] | 0.84 [0.72 to 0.92]
  B/Yamagata Visit 4 GMFR ≥ 4-Fold Rise: number analyzed (Participants) | 57 | 56
  B/Yamagata Visit 4 GMFR ≥ 4-Fold Rise | 0.09 [0.03 to 0.19] | 0.22 [0.12 to 0.35]

3. Secondary Outcome: Solicited Local Injection Site Adverse Events
Description: The proportion of subjects in each group experiencing at least one solicited AE with 95% posterior credible intervals, separated by vaccine number and adverse event type. AEs were assessed by clinicians using Tables 4 and 5 within section C16 of the protocol.
  Solicited injection site AEs included: pain, tenderness, erythema/redness, and swelling/induration. The diameter of any erythema/redness and swelling/induration was measured to evaluate "redness size" and "swelling size."
Time Frame: Adverse events were recorded for 7 days following each vaccination or until resolution, up to study conclusion.
Population: The number of subjects analyzed for Vaccine 1 represents the number of subjects who attended Visit 1 and received the first vaccine. The number of subjects analyzed for Vaccine 2 represents the number of subjects who attended Visit 2 and received the second vaccine.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Number analyzed (Participants) | 60 | 64
proportion of participants
  Vaccine 1 - Pain | 0.250 [0.147 to 0.379] | 0.156 [0.078 to 0.269]
  Vaccine 1 - Tenderness | 0.383 [0.261 to 0.518] | 0.297 [0.189 to 0.424]
  Vaccine 1 - Redness size | 0.067 [0.018 to 0.162] | 0.047 [0.010 to 0.131]
  Vaccine 1 - Swelling | 0.117 [0.048 to 0.226] | 0.094 [0.035 to 0.193]
  Vaccine 1 - Swelling size | 0.100 [0.038 to 0.205] | 0.063 [0.017 to 0.152]
  Vaccine 2 - Pain: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Pain | 0.254 [0.150 to 0.384] | 0.169 [0.084 to 0.290]
  Vaccine 2 - Tenderness: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Tenderness | 0.458 [0.327 to 0.592] | 0.288 [0.178 to 0.421]
  Vaccine 2 - Redness size: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Redness size | 0.102 [0.038 to 0.208] | 0.000 [0.000 to 0.061]
  Vaccine 2 - Swelling: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Swelling | 0.136 [0.060 to 0.250] | 0.102 [0.038 to 0.208]
  Vaccine 2 - Swelling size: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Swelling size | 0.119 [0.049 to 0.229] | 0.034 [0.004 to 0.117]

4. Secondary Outcome: Solicited Systemic Adverse Events
Description: The proportion of subjects in each group experiencing at least one solicited AE with 95% posterior credible intervals, separated by vaccine number and adverse event type. AEs were assessed by clinicians using Tables 4 and 5 within section C16 of the protocol.
  Solicited systemic AEs included: fevers, fatigue/malaise, headache, nausea, body ache/myalgia, generally activity, and vomiting.
Time Frame: Adverse events were recorded for 7 days following each vaccination or until resolution, up to study conclusion.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Number analyzed (Participants) | 60 | 64
proportion of participants
  Vaccine 1 - Fever | 0.033 [0.004 to 0.115] | 0.031 [0.004 to 0.108]
  Vaccine 1 - Fatigue | 0.350 [0.231 to 0.484] | 0.313 [0.202 to 0.441]
  Vaccine 1 - Headache | 0.267 [0.161 to 0.397] | 0.188 [0.101 to 0.305]
  Vaccine 1 - Nausea | 0.083 [0.028 to 0.184] | 0.172 [0.089 to 0.287]
  Vaccine 1 - Myalgia | 0.200 [0.108 to 0.323] | 0.172 [0.089 to 0.287]
  Vaccine 1 - General Activity | 0.300 [0.188 to 0.432] | 0.297 [0.189 to 0.424]
  Vaccine 1 - Vomiting | 0.017 [0.000 to 0.089] | 0.063 [0.017 to 0.152]
  Vaccine 2 - Fever: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Fever | 0.034 [0.004 to 0.117] | 0.068 [0.019 to 0.165]
  Vaccine 2 - Fatigue: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Fatigue | 0.254 [0.150 to 0.384] | 0.254 [0.150 to 0.384]
  Vaccine 2 - Headache: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Headache | 0.203 [0.110 to 0.328] | 0.203 [0.110 to 0.328]
  Vaccine 2 - Nausea: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Nausea | 0.119 [0.049 to 0.229] | 0.186 [0.097 to 0.309]
  Vaccine 2 - Myalgia: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Myalgia | 0.153 [0.072 to 0.270] | 0.153 [0.072 to 0.270]
  Vaccine 2 - General Activity: number analyzed (Participants) | 59 | 59
  Vaccine 2 - General Activity | 0.305 [0.192 to 0.439] | 0.220 [0.123 to 0.347]
  Vaccine 2 - Vomiting: number analyzed (Participants) | 59 | 59
  Vaccine 2 - Vomiting | 0.000 [0.000 to 0.061] | 0.017 [0.000 to 0.091]

5. Secondary Outcome: Percentage of Individuals in Each Group That Test Positive for Influenza by PCR
Description: The percentage of breakthrough flu in vaccinated participants, separated by treatment group.
Time Frame: Nasal swabs were collected at each study visit or within 48 hours if a subject presented with influenza-like symptoms throughout the duration of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
Number analyzed (Participants) | 60 | 64
Participants | 5 | 2

6. Other Pre Specified Outcome: B Cell Response Assessed by Mass Cytometry and In-vitro Functionality Assays
Description: The total number of B cells will be measured prior to each vaccination and compared to each group.
Time Frame: Visit 1 cell counts (baseline) were measured on day 0; visit 2 cell counts were measured 28-42 days after visit 1; visit 3 cell counts were measured 28-42 days after visit 2; and visit 4 cell counts were measured 138-222 days after visit 2.
Reporting Status: Not Posted, anticipated posting 2025-08

7. Other Pre Specified Outcome: T Cell Response Assessed by Mass Cytometry and In-vitro Functionality Assays
Description: The total number of T cells will be measured prior to each vaccination and compared to each group.
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for 7 days following each vaccination (up to day 7 for vaccine 1 and up to day 35-49 for vaccine 2). Events were followed until resolution, up to study conclusion.
Arm/Group | Group I (HD-TIV) | Group 2 (SD-QIV)
All-Cause Mortality (participants affected / at risk) | 2/60 | 5/64
Serious Adverse Events (participants affected / at risk) | 4/60 | 0/64
Other Adverse Events (participants affected / at risk) | 45/60 | 45/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (HD-TIV) (N=60) | Group 2 (SD-QIV) (N=64)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Viral illness (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (HD-TIV) (N=60) | Group 2 (SD-QIV) (N=64)
Fever (General disorders) | 4 (4) | 6 (6) — Temperature of 100.4 degrees Fahrenheit or greater Systemic solicited reaction
Fatigue (General disorders) | 24 (24) | 23 (23) — Systemic solicited reaction
Headache (General disorders) | 18 (18) | 20 (20) — Systemic solicited reaction
Nausea (General disorders) | 10 (10) | 16 (16) — Systemic solicited reaction
Myalgia/ Body aches (General disorders) | 15 (15) | 18 (18) — Systemic solicited reaction
Decreased general activity (General disorders) | 26 (26) | 25 (25) — Systemic solicited reaction
Vomiting (General disorders) | 1 (1) | 5 (5) — Systemic solicited reaction
Pain (General disorders) | 21 (21) | 15 (15) — Solicited injection-site reaction
Tenderness (General disorders) | 33 (33) | 23 (23) — Solicited injection-site reaction
Swelling (Skin and subcutaneous tissue disorders) | 11 (11) | 9 (9) — Solicited injection-site reaction
Redness/ Erythema (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) — Injection-site reaction of at least 0.5 cm in diameter Solicited injection-site reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03179761/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03179761/ICF_001.pdf